CLINICAL TRIAL: NCT02457754
Title: Physical Fitness and Bone Structure Evaluation in Preschool Children
Status: Completed | Type: Observational
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, German Vicente-Rodríguez, Dr., Universidad de Zaragoza
Other Study IDs: JIUZ-2014-BIO-08-216-162
Record Dates: First submitted 2015-03-20; First posted 2015-05-29 (Estimated); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Child, Preschool; Bone Structure; Physical Fitness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
Several studies have shown a high association between physical fitness and present and future health. Two of the main epidemics of the industrialized world are obesity and osteoporosis, diseases that could be prevented with early interventions from childhood. Both, physical activity and physical fitness have shown an association with these diseases, but tools for assessing them in early ages are still in development. Moreover, there is a lack of physical fitness reference values in preschool children and the relation of pathologies with physical fitness in these ages is still to be demonstrated. Therefore, through a simple and precise methodology displayed in the school and adapted for the younger we intend to: Provide a combination of safe and precise field tests to evaluate health related physical fitness in preschool children. Analyze body composition, risk of overweight, obesity and low mineral density and their relation with physical activity. The evaluation of these health-related physical fitness variables in early ages is of great interest to clinic and public health.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* 3 to 5 years old

Exclusion Criteria:

* Unhealthy
* Taking drugs affecting bone

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy 3 to 5 year-old children
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Assessment of physical fitness in preschool children | 4 months evaluation

CONTACTS AND LOCATIONS:
Overall Officials: German Vicente-Rodríguez, PhD, Principal Investigator — Universidad de Zaragoza
Locations (1):
- Universidad de Zaragoza, Zaragoza, Spain